CLINICAL TRIAL: NCT06451965
Title: A Single Case Experiment Design Investigating Wisdom Enhancement to Augment CBT Outcomes for Depression in Post-Stroke Populations
Brief Title: SCED - Wisdom Enhancement for Post-Stroke Depression
Acronym: WE-PSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 335191
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-05

CONDITIONS: Post-stroke Depression
Keywords: wisdom; CBT; cognitive behavioural therapy; stroke; depression
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Wisdom Enhancement Timeline Intervention (Experimental): Participants first complete a baseline observation phase of 2, 3, or 4 weeks (duration randomly assigned). During this phase, no intervention is provided and daily visual analogue scale ratings are recorded, along with administration of the PHQ-9 at the start of the phase. The baseline phase is then followed by six weekly one-hour therapy sessions delivering the Wisdom Enhancement Timeline intervention, during which daily ratings continued and the PHQ-9 was administered again at the end.
  Interventions: Other: Timeline Intervention

INTERVENTIONS:
Other: Timeline Intervention — The proposed intervention consists of six sessions. In Session One, the focus is on building rapport, assessing individual difficulties, setting client-focused goals, and introducing the timeline. Participants complete timeline examples during the session and as homework.
  In Session Two, psychoeducation is provided regarding the impact of stroke, addressing changes in identity and associated feelings of grievance.
  Session Three onwards introduces active change methods, encouraging reflection on complex life events. The aim is to promote resilience, meaning, self-compassion, and self-acceptance by exploring past coping strategies and finding significance in events of regret. This framework aims to enhance research on complex interventions, considering efficacy, effectiveness, theory-based approaches, and systems perspectives.

SUMMARY:
One-third of stroke survivors experience post-stroke depression, but there are currently no official guidelines for supporting them. Researchers aim to investigate whether the wisdom enhancement timeline technique can reduce depression in stroke survivors. The investigators also want to understand how this technique positively impacts mood, identity, self-esteem, and wisdom. The study will involve nine stroke survivors from the National Health Service (NHS) to gain insights into effective ways to support those with post-stroke depression.

DETAILED DESCRIPTION:
One-third of stroke survivors have post-stroke depression. Finding ways to help them feel more positive after such a challenging event can be tricky. Right now, there are no official guidelines on the best way to support post-stroke depression, and research into this is still growing. That is why the investigators want to see if the wisdom enhancement timeline can improve the mood and overall well-being of people who have had a stroke.

In this study, the investigators have two goals. First, the investigators want to see if the wisdom enhancement timeline technique can reduce depression in stroke survivors. Second, the investigators aim to discover how this technique brings positive mood changes.

The main question the investigators want to answer

1. Does enhancing wisdom through the timeline technique improve psychological outcomes (mood, identity, self-esteem) in post-stroke depressed individuals?
2. In post-stroke depressed individuals, is the improvement in wisdom the first indicator of subsequent improvements in identity, self-esteem, and mood?

It is hypothesised that wisdom will improve first following the session where wisdom is applied. This will then be followed by either identity or self-esteem, with mood improving last.

To carry out this study, the investigators will work with three stroke survivors receiving care from the National Health Service (NHS). By focusing on this smaller group, the investigators hope to gain insights into the effectiveness of the technique in reducing depression and enhancing the lives of stroke survivors. This study is essential as it could help the investigators understand the best way to support those with post-stroke depression.

ELIGIBILITY:
Inclusion Criteria:

* Had a stroke.
* Those who self-report as having difficulties with depression to a clinician.
* Have sufficient cognitive and communication abilities for informed consent and active engagement

Exclusion Criteria:

* Under the age of 18. Because this is the age when they are treated as an adult by UK law.
* Severe cognitive impairments or mental health difficulties that would hinder task engagement or provide informed consent.
* Medical instability jeopardising consistent participation or well-being.
* Significant risk concerns regarding safety to themselves or others.
* Substance use/dependency impacting adherence.
* Prescribed psychotropic medication less than 3 months ago.
* Currently involved in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ercan T Hassan, PGDIP CBT, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following submission of the thesis, the entire documentation will be stored on the universities repository.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: All information will be kept on the University of East Anglia's repository. This will remain there for 10 years. All participant information will be anonymised to protect their confidentiality.
Access Criteria: No criteria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via a local NHS Stroke service. 3 consented to participate in the trial with all completing it.
Pre-assignment Details: No participants were excluded.
Period: Overall Study
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
Started | 3
Baseline Phase - 2 Weeks | 1
Baseline Phase - 3 Weeks | 1
Baseline Phase - 4 Weeks | 1
Intervention Phase | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — Age at enrollment
  Participants
    <=18 years | 0
    Between 18 and 65 years | 2
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported sex at enrollment.
  Participants
    Female | 2
    Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
PHQ-9 Score at Baseline [Mean (Standard Deviation); unit: Score 0-27] — Patient Health Questionnaire-9 total score, range 0-27; higher scores indicate more severe depressive symptoms.
  Score 0-27 | 16.33 (4.62)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) - Mood
Description: A single-item Visual Analogue Scale was used to assess mood, rated daily on a 0-10 scale, where 0 indicates "worst possible mood" and 10 indicates "best possible mood." Three participants recorded their rating once each day throughout the trial.
Time Frame: Daily during baseline phase and intervention phase (total of 8-10 weeks depending on baseline length)
Population: All three participants who started the study were included in the analysis. Daily visual analogue scale ratings for mood (0-10) were collected throughout each participant's baseline and intervention phases. The values reported in the table represent the mean (SD) of all daily ratings across each phase for all participants. No participants were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
Number analyzed (Participants) | 3
Scores on a scale
  Baseline phase (mean across participants) | 3.53 (0.81)
  Intervention phase (mean across participants) | 5.23 (1.85)

2. Primary Outcome: Visual Analogue Scale (VAS) - Identity
Description: A single-item Visual Analogue Scale was used to assess identity, rated daily on a 0-10 scale, where 0 indicates "a disconnect from who they are" and 10 indicates "complete connection." Three participants recorded their rating once each day throughout the baseline and intervention phases.
Time Frame: Daily during baseline phase and intervention phase (total of 8-10 weeks depending on baseline length)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
Number analyzed (Participants) | 3
Scores on a scale
  Baseline phase (mean across participants) | 2.55 (1.21)
  Intervention phase (mean across participants) | 5.09 (2.33)

3. Primary Outcome: Visual Analogue Scale (VAS) - Wisdom
Description: A single-item Visual Analogue Scale was used to assess Wisdom, rated daily on a 0-10 scale, where 0 indicates "low wisdom" and 10 indicates "high wisdom." Participants recorded their rating once each day throughout the baseline and intervention phases.
Time Frame: Daily during baseline phase and intervention phase (total of 8-10 weeks depending on baseline length)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
Number analyzed (Participants) | 3
Scores on a scale
  Baseline phase (mean across participants) | 2.79 (1.33)
  Intervention phase (mean across participants) | 5.56 (2.08)

4. Primary Outcome: Visual Analogue Scale (VAS) - Self-esteem
Description: A single-item Visual Analogue Scale was used to assess self-esteem, rated daily on a 0-10 scale, where 0 indicates "low self-esteem" and 10 indicates "high self-esteem." Participants recorded their rating once each day throughout the baseline and intervention phases.
Time Frame: Daily during baseline phase and intervention phase (total of 8-10 weeks depending on baseline length)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
Number analyzed (Participants) | 3
Scores on a scale
  Baseline phase (mean across participants) | 3 (0.96)
  Intervention phase (mean across participants) | 4.92 (2.01)

5. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a 9-item self-report measure assessing the severity of depressive symptoms over the past two weeks. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), producing a total score between 0 and 27, with higher scores indicating more severe depression.
Time Frame: Baseline to end of 6-week intervention phase
Population: All three participants who started the study were included in the analysis. The PHQ-9 was administered at the start of the baseline phase (week 0, pre-intervention) and again at the end of the intervention phase (week 8-10, depending on baseline duration). The values reported in the table represent the mean (SD) of participants' total scores at these time points. No participants were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
Number analyzed (Participants) | 3
Scores on a scale
  Baseline (week 0, pre-intervention) | 13.66 (4.61)
  Post-intervention (week 8-10) | 7.33 (1.15)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: All participants (n=3) were monitored for adverse events via non-systematic self-report and clinician observation throughout the 10-week study period. No deaths, serious adverse events, or other adverse events were observed. No deviations from ClinicalTrials.gov definitions were made.
Arm/Group | Experimental: Wisdom Enhancement Timeline Intervention
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT06451965/Prot_SAP_000.pdf